CLINICAL TRIAL: NCT01895517
Title: Randomized Controlled Trial to Evaluate the Efficacy of Concurrent Liquid-based Cytology ( LBC) and HPV DNA Testing Versus LBC Alone for the Primary Cervical Cancer Screening
Brief Title: CervIcal Cancer Screening Trial by Randomization of HPV Testing Intervention for Upcoming Screening （CITRUS Study）
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Translational Research Center for Medical Innovation, Kobe, Hyogo, Japan (Other)
Collaborators: Keio University (Other); Jikei University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: TRIUC1312; UMIN000010843 (Registry Identifier: UMIN Clinical Trials Registry (UMIN-CTR))
Record Dates: First submitted 2013-07-04; First posted 2013-07-10 (Estimated); Last update posted 2023-06-26 (Actual); Status verified 2022-05

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — AKAP13 protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LBC (Active Comparator): Cervical cancer screening by using liquid based cytology as a standard screening modality
  Interventions: Other: LBC
- LBC plus HPV DNA testing (Experimental): Cervical cancer screening by using liquid based cytology plus HPV DNA testing as an experimentally screening modality
  Interventions: Other: LBC plus HPV DNA testing

INTERVENTIONS:
Other: LBC — Cervical cancer screening by using liquid based cytology as a standard screening modality
  Arms: LBC
Other: LBC plus HPV DNA testing — Cervical cancer screening by using liquid based cytology plus HPV DNA testing as an experimentally screening modality
  Arms: LBC plus HPV DNA testing

SUMMARY:
The aim of this study is to assess efficacy of the screening with concurrent liquid-based cytology and HPV DNA testing for the primary cervical cancer screening over 7 years.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 30-64 years old
2. Participants provided written informed consent

Exclusion Criteria:

Women who

1. will receive planed HPV DNA testing by local governmental cervical cancer program next six years
2. have had cervical invasive cancer before
3. have undergone cervical conization
4. have undergone hysterectomy
5. have had or have the cytological abnormalities and are under follow-up
6. are pregnant
7. are judged ineligible for this trial by physician

Ages: 30 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18471 (Actual)
Dates: Start 2013-06-07 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
The incidence of cervical intraepithelial neoplasia(CIN)3 or worse during the whole period | 6 years

SECONDARY OUTCOMES:
The incidence of CIN3 or worse at baseline, and two years, four years, and six years post baseline | 2 years, 4 years, 6 years
The incidence of CIN2 or worse at baseline, and two years, four years, and six years post baseline | 2 years, 4 years, 6 years
The incidence of CIN1 or worse at baseline, and two years, four years, and six years post baseline | 2 years, 4 years, 6 years
The incidence of invasive cancer at baseline, and two years, four years, and six years post baseline | 2 years, 4 years, 6 years
The number of cervical cytology performance | 6 years
The number of colposcopy and biopsy performance | 6 years

CONTACTS AND LOCATIONS:
Locations (1):
- School of Medicine, Keio University, Shinjuku, Tokyo, Japan

REFERENCES:
- [Derived] Morisada T, Teramoto K, Takano H, Sakamoto I, Nishio H, Iwata T, Hashi A, Katoh R, Okamoto A, Sasaki H, Nakatani E, Teramukai S, Aoki D. CITRUS, cervical cancer screening trial by randomization of HPV testing intervention for upcoming screening: Design, methods and baseline data of 18,471 women. Cancer Epidemiol. 2017 Oct;50(Pt A):60-67. doi: 10.1016/j.canep.2017.07.017. Epub 2017 Aug 16. PMID 28818742